CLINICAL TRIAL: NCT05025735
Title: Alpelisib, Fulvestrant and Dapagliflozin for the Treatment of HR+, HER2 -, PIK3CA Mutant Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saint Luke's Health System (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBYL719A0US03T
Record Dates: First submitted 2021-06-26; First posted 2021-08-27 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Metastatic Breast Cancer; HER2-negative Breast Cancer
Keywords: Metastatic Breast Cancer; HER2 Negative; HR Positive
MeSH Terms: conditions — Breast Neoplasms | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: open label pilot to test the combination of dapagliflozin, a commercially available SGLT-2 inhibitor, in combination with alpelisib + fulvestrant in patients with HR+/HER2- mBC.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Phase 2 study of Fulvestrant, alpelisib and dapagliflozin (Experimental): A cycle length is defined as 28 days.
  Fulvestrant 500 mg intramuscular, Cycle 1, Day 1 and Day 15; Cycle 2 and beyond 500 mg Intramuscular Day 1.
  Alpelisib 300 mg by mouth, daily, continuously beginning on Cycle 1, Day 1.
  Dapagliflozin 10 mg by mouth, daily, continuously beginning Cycle 1, Day 3.
  Interventions: Drug: Dapagliflozin 10Mg Tab

INTERVENTIONS:
Drug: Dapagliflozin 10Mg Tab — Hyperglycemia is an expected effect of PI3K inhibitors given the pivotal role of PI3K in mediating the response to insulin in multiple tissues. Blocking insulin signaling by p110α inhibitors leads to glycogen breakdown in the liver along with decreased glucose uptake in peripheral tissues. The resulting hyperglycemia causes a compensatory response of increase insulin secretion by the pancreas.
  If concurrent treatment with dapagliflozin can abrogate the alpelisib induced hyperglycemia and subsequent rebound hyperinsulinemia it may significantly improve the therapeutic efficacy of alpelisib.

SUMMARY:
This will be a single arm, open label pilot to test the combination of dapagliflozin, a commercially available SGLT-2 inhibitor, in combination with alpelisib + fulvestrant in patients with HR+/HER2- mBC. The objective of this study is to determine if the addition of dapagliflozin to the combination of alpelisib and fulvestrant leads to significant reduction in all-grade hyperglycemia.

DETAILED DESCRIPTION:
Alpelisib is a p110α specific PI3K inhibitor that has shown significant clinical benefit in patients with HR+/HER2 negative mBC harboring activating PIK3CA mutations. The SOLAR-1 study randomized patients with MBC progressing after aromatase inhibitor therapy patients had a PFS of 11 months with fulvestrant plus alpelisib versus 5.7 months with fulvestrant alone. Alpelisib was associated with a 65% incidence of hyperglycemia, including 37% Grade 3 or 4 hyperglycemia.

Hyperglycemia is an expected effect of PI3K inhibitors given the pivotal role of PI3K in mediating the response to insulin in multiple tissues. Blocking insulin signaling by p110α inhibitors leads to glycogen breakdown in the liver along with decreased glucose uptake in peripheral tissues. The resulting hyperglycemia causes a compensatory response of increase insulin secretion by the pancreas.

Cantley and colleagues have shown in animal models that treatment with BYL-719(alpelisib) results in rapid increase in plasma glucose level and a compensatory increase in insulin.

They went on to show that this rebound hyperinsulinemia was able to rescue KPC tumor allografts from BYL-719 inhibition as evidenced by increasing phosphorylation of downstream effectors in the PI3K pathway, pAKT and PS6. Pretreatment of the mice with an SGLT-2 inhibitor decreased the hyperglycemia and hyperinsulinemia following treatment with BYL-719. Importantly, the response of the KPC tumor allografts to treatment was concordant with reduction in insulin levels.3

This provides a rationale for combining dapagliflozin with alpelisib in the treatment of HR+, PIK3CA mutant MBC. If concurrent treatment with dapagliflozin can abrogate the alpelisib induced hyperglycemia and subsequent rebound hyperinsulinemia it may significantly improve the therapeutic efficacy of alpelisib.

ELIGIBILITY:
Inclusion Criteria:

1. Patients > 18 years old with stage IV or locally advanced, unresectable Stage III breast cancer that is:

   1. ER and/or PR positive by local laboratory evaluation
   2. HER2 negative as defined by: either IHC status of 0, 1+ ; IHC of 2+ with FISH negative by ASCO/CAP guidelines.
2. If female, post-menopausal status as defined by

   1. Prior bilateral oophorectomy
   2. Age > 60
   3. Age <60 and amenorrheic for 12 or more months in the absence of chemotherapy, tamoxifen, toremifene; or ovarian suppression and Follicle-stimulating Hormone (FSH) and estradiol in the postmenopausal range per local normal range.
   4. Current use of LHRH agonist for ovarian suppression and estradiol and FSH documented in the post-menopausal range.
3. PIK3CA activating mutation identified by a either in a CLIA certified tumor genomic assay or ctDNA assay.
4. Patients may be:

   1. relapsed with documented evidence of progression while on (neo) adjuvant endocrine therapy or within 12 months from completion of (neo)adjuvant endocrine therapy with no treatment for metastatic disease
   2. relapsed with documented evidence of progression more than 12 months following/completion of (neo)adjuvant endocrine therapy and then subsequently progressed with documented evidence of progression while on or after only one line of endocrine therapy for metastatic disease
   3. newly diagnosed advanced breast cancer, then relapsed with documented evidence of progression while on or after only one line of endocrine therapy
   4. Prior endocrine treatment must have included a CDK4/6 inhibitor
5. ECOG performance status 0-2
6. Patient has adequate bone marrow and organ function as defined by the following laboratory values:

   1. Absolute neutrophil count ≥ 1.0 × 109/L
   2. Platelets ≥ 75 × 109/L
   3. Hemoglobin ≥ 8.0 g/dL
   4. Calcium (corrected for serum albumin) and magnesium within normal limits or ≤ grade 1 according to NCI-CTCAE version 4.03 if judged clinically not significant by the investigator
   5. Potassium within normal limits, or corrected with supplements
   6. Creatinine Clearance 35 ≥ mL/min using Cockcroft-Gault formula
   7. In absence of liver metastases, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3.0 × ULN. If the patient has liver metastases, ALT and AST ≤ 5 × ULN
   8. Total bilirubin < ULN except for patients with Gilbert's syndrome who may only be included if the total bilirubin is ≤ 3.0 × ULN or direct bilirubin ≤ 1.5 × ULN≤
7. Fasting plasma glucose (FPG) ≤ 200 and Glycosylated Hemoglobin (HbA1c) ≤ 6.5%
8. Fasting Serum amylase ≤ 2 × ULN
9. Fasting Serum lipase ≤ ULN

Exclusion Criteria:

1. Patient has not recovered from all toxicities related to prior anticancer therapies to NCI CTCAE version 4.03 Grade ≤1. Exception to this criterion: patients with any grade of alopecia are allowed to enter the study.
2. Patient with symptomatic visceral disease or any disease burden that makes the patient ineligible for endocrine therapy per the investigator's best judgment.
3. Patients with Type I diabetes or history of diabetic ketoacidosis
4. Patient has received prior treatment with chemotherapy in the metastatic setting, fulvestrant, any PI3K, mTOR or AKT inhibitor
5. Patient has a known hypersensitivity to alpelisib or fulvestrant, or to any of the excipients of alpelisib or fulvestrant.
6. Patient is concurrently using other anti-cancer therapy.
7. Patient has had surgery within 14 days prior to starting study drug or has not recovered from major side effects of surgery.
8. Patient has central nervous system (CNS) involvement that does not meet ALL of the following criteria:

   * completed prior therapy (including radiation and/or surgery) for CNS metastases ≥ 14 days prior to the start of study and
   * CNS tumor is clinically stable at the time of screening and
   * patient is not receiving steroids and/or enzyme inducing anti-epileptic medications for brain metastases
9. Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
10. Patient is following a ketogenic diet and unwilling to change diet.
11. Patient has any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, contraindicate patient participation in the clinical study.
12. Patient has currently documented pneumonitis (the chest CT scan performed at baseline for the purpose of tumor assessment should be reviewed to confirm that there are no relevant pulmonary complications present).
13. Patient is currently receiving or has received systemic corticosteroids 7 days prior to starting study drug, or who have not fully recovered from side effects of such treatment.

    Note: The following uses of corticosteroids are permitted: single doses, topical applications (e.g., for rash), inhaled sprays (e.g., for obstructive airways diseases), eye drops or local injections (e.g., intra-articular).
14. Sexually active males unless they are sterilized (at least 6 months prior to screening) or use a condom during intercourse while taking drug and for at least 8 months after stopping alpelisib and/or fulvestrant. .
15. Participation in a prior investigational study within 14 days prior to the start of study treatment or within 5 half-lives of the investigational product, whichever is longer.
16. Not able to understand and to comply with study instructions and requirements.
17. History of acute pancreatitis within1 year of screening or past medical history of chronic pancreatitis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-08-25 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of all grade hyperglycemia as assessed by CTCAE v5.0 | Through study completion, an average of 1 year.

SECONDARY OUTCOMES:
Incidence of Grade 3/4 hyperglycemia as assessed by CTCAE v5.0 | Through study completion, an average of 1 year.
Overall response rate (ORR) as assed by RECIST 1.1 in patients with measurable disease | Through study completion, an average of 1 year.
Progression free survival | Through study completion, an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J Pluard, MD, Principal Investigator — Saint Luke's Cancer Institute
Locations (1):
- Saint Luke's Cancer Institute, Kansas City, Missouri, United States